CLINICAL TRIAL: NCT01363193
Title: Assessing Safety and Efficacy of Lean Body Weight-based Intravenous Heparin Dosing in Obese/Morbidly Obese Patients. A Pilot Study
Brief Title: Safety and Efficacy of Lean Body Weight-based IV Heparin Dosing in Obese/Morbidly Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nazareth Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBW Heparin study
Record Dates: First submitted 2011-04-25; First posted 2011-06-01 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Obesity; Morbid Obesity; Venous Thromboembolism; Atrial Fibrillation; Angina; Chest Pain
Keywords: Weight-based heparin dosing; Obesity; Body Mass Index; Venous thromboembolism; Atrial fibrillation; Lean body weight; Unfractionated heparin; heparin
MeSH Terms: conditions — Obesity; Obesity, Morbid; Venous Thromboembolism; Atrial Fibrillation; Angina Pectoris; Chest Pain | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lean Body Weight-based heparin dose — For patients who meet the inclusion criteria including body mass index of 30 and greater (and do not have any exclusion criteria), will have intravenous weight-based heparin (unfractionated heparin) dose based on their Lean body weight.
  Lean Body Weight is based on the formula by Janmahasatian et al. 2005. Calculated by a computer program; Male = [9270 x weight (kg)] / [6680+216 x BMI] Female = [9270 x weight (kg)] / [8780+244 x BMI]
  Other Names: unfractionated heparin

SUMMARY:
Standard weight-based IV heparin for normal weight patients is based on actual body weight (ABW). However, no well-defined guidelines have been established for patients considered to be obese or morbidly obese. In current practice, the calculated ABW based heparin initial bolus dose and infusion rates are quite high, and therefore often not used for obese/morbidly obese patients for fear of bleeding.

Heparin is distributed in the body approximately the same as blood and does not get distributed to adipose tissue. There are some studies suggesting that lean body weight (LBW) might be a better basis for dosing heparin. LBW is a calculated weight that excludes the weight of fat.

The investigators hypothesize that intravenous heparin dosing based on the Lean body weight of obese/morbidly obese patients would be safe and effective in achieving a therapeutic level of heparin in 24 hours compared to the usual practice in this patient population.

DETAILED DESCRIPTION:
Unfractionated Heparin has been used as an anticoagulant in various disease states and conditions, such as atrial fibrillation, deep vein thrombosis (DVT), pulmonary embolism (PE), myocardial infarction, acute coronary syndrome, and peripheral vascular disease. Prior studies have demonstrated that a weight-based heparin (WBH) dosing regimen is superior to a fixed dosing regimen (e.g. 5000 units bolus and 1000 units/hour) in achieving a therapeutic activated partial thromboplastin time (aPTT) more quickly and with fewer complications (1,2). The importance of achieving anticoagulation to a targeted aPTT range within 24 hours after starting intravenous heparin infusion has demonstrated a therapeutic benefit (1,3,30-31). WBH dosing is now the standard of care for intravenous heparin therapy.

Prior studies have assessed the benefit of WBH utilizing the patients' actual body weight (ABW), but have not significantly considered the issue of dosing and titrating WBH in the obese and morbidly obese (O/MO) patient population (1,16-17, 32). There are few studies that have examined the effect of obesity in heparin dosing, and there are wide variations in how obesity is defined and how (if at all) WBH nomograms based on ABW are adjusted in this patient population (4,12,16-18, 23, 25). In addition, there are but a few case reports addressing WBH-dosing in the O/MO patient population according to a more modern definition of obesity. These limitations make it difficult to apply in the clinical setting (16-18, 21-28). In current practice, ABW-based heparin bolus doses and infusion rates are quite high and therefore often not used for O/MO patients due to fears of over-anticoagulation and of serious bleeding. Studies have in fact reported a higher potential of supratherapeutic aPTT in the bariatrically-challenged population (19, 23-24, 26-27). Therefore, it remains uncertain as to how to optimize intravenous heparin dosing in these patients.

The volume of distribution (Vd) of heparin is similar to blood volume and adipose tissue has little vasculature to account for heparin's distribution (5-11). LBW has recently been proposed to be a better metric for dosing heparin in obese/morbidly obese patients (14-15,20,29,34).

The investigators hypothesize that intravenous heparin (IVH) dosing based on LBW of O/MO patients would be safe and effective in achieving aPTT within 24 hours compared to the usual practice in this patient population. In addition, the investigators postulate that it would be cost-effective since it would reduce the number of blood draws and laboratory tests (13).

This prospective study will involve the departments of emergency medicine, internal medicine (sections of cardiology and critical care), laboratory, nursing, and pharmacy. Those patients who are O/MO according to 2004 World Health Organization (WHO) definition (BMI > 30) (33) and have an IVH order will be enrolled to receive heparin via a LBW-based nomogram.

As a comparison, the investigators will also have the calculated initial bolus and infusion doses that would have been given in a traditional ABW-based treatment algorithm.

A signed consent form from the patients will be obtained in order to use the LBW-based heparin nomogram. In accordance with the standard weight-based heparin protocol and 2008 CHEST guidelines, the modified version of current Mercy Nazareth Hospital (MNH) weight-based heparin protocol will be followed in all other aspects beyond the dosing nomogram. An aPTT tracking form and data collection tool will be utilized to monitor and gather results.

References on File - provided upon request.

ELIGIBILITY:
Inclusion Criteria:

* Patients with body mass index greater than or equal to 30
* Patients admitted to Nazareth Hospital inpatient units
* Weight-based intravenous heparin, with a diagnosis of atrial fibrillation, suspected or confirmed deep vein thrombosis or pulmonary embolism, unstable angina or Non ST elevation myocardial infarction with hemodynamic stability, or peripheral vascular disease, ordered at the time of admission/transfer or during the patient stay in the Intensive Care unit or Progressive Care unit.
* Prior permission from the patient's attending physician
* Permission from the physician who ordered the intravenous weight-based heparin (if different from the attending)
* Signed consent form by the patient.

Exclusion Criteria:

* Patients with stroke, TIA, or ST elevation myocardial infarction
* Patients who have hemodynamic or cardiopulmonary instability at the time of intravenous heparin order
* Patients with thrombophilia
* Patients who are pregnant or may be pregnant
* Those patients who have been on any oral anticoagulants (Warfarin, rivaroxaban, dabigatran or apixaban), treatment dose of other anticoagulants or intravenous thrombolytics in previous 7 days.
* Patients who have a PTT greater than 37 seconds.
* History of heparin-induced thrombocytopenia or known allergy to heparin
* Deviation from the Weight-based heparin protocol ordered by a physician at the time intravenous heparin was written (i.e. no bolus dose ordered, different target therapeutic aPTT range, different bolus dose per kg, etc.)
* Informed consent either refused or not obtained
* Objection from a physician caring for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Percent of study patients achieving therapeutic aPTT within first 24 hours on a hospital based IV heparin protocol using Lean Body Weight | 24 hours

SECONDARY OUTCOMES:
Evaluation of side effects and/or complications during the index hospitalization | participants will be followed for the duration of hospital stay, usually 7 days or less
  Evaluation of side effects/complications - bleeding, other events related to heparin therapy such as Heparin-induced thrombocytopenia and recurrent thromboembolism during study period.
  Study duration/completion - until discontinuation of heparin or discharge from inpatient hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel J Park, PharmD, BCPS, Principal Investigator — Nazareh Hospital - Mercy Health System
Locations (1):
- Nazareth Hospital - Mercy Health System, Philadelphia, Pennsylvania, United States